CLINICAL TRIAL: NCT06231784
Title: Prospective, Open-label Clinical Study to Evaluate the Efficacy and Function of the AkkoLens Accommodative Intraocular Acrylic Lens for the Treatment of Cataracts
Brief Title: Efficacy of the AkkoLens IOL in Patients With Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Collaborators: AkkoLens Clinical bv (Unknown)
Responsible Party: Principal Investigator, Jorge Alio, Dr, Vissum, Instituto Oftalmológico de Alicante
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lumina
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cataract
Keywords: Intraocular lens; Accommodation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: LUMINA IOL
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumina Implantation (Other): Patients implanted with LUMINA IOL
  Interventions: Device: LUMINA IOL

INTERVENTIONS:
Device: LUMINA IOL — A standard technique of phacoemulsification was performed followed by implantation of the Lumina in the sulcus plane of the eye by using a standard disposable injector system with an adapted, proprietary, AkkoLens butterfly cartridge.

SUMMARY:
The goal of this observational study is to learn about the verification of the effectiveness and visual acuity of LUMINA in patients after lens replacement due to cataracts.

The main questions it aims to answer are:

* Evaluation of the effectiveness of the LUMINA lens in patients after lens replacement due to cataracts
* Evaluation of the accommodative power of the LUMINA lens. Participants will have cataract surgery and the IOL LUMINA will be implanted in the sulcus.

DETAILED DESCRIPTION:
This is an observational, prospective, longitudinal, and consecutive study involving patients with clinical cataract eligible for cataract surgery who opt for the implantation of the Lumina (Akkolens, Clinical BV, The Netherlands) accommodative lens. The study was conducted at the Cornea, Cataract, and Refractive Surgery Unit in Vissum Alicante, Miranza Group, Spain. The study adhered to the tenets of the Declaration of Helsinki (2013 version )and was approved by the Comite Etico de Investigacion Clinica Vissum Alicante.

The study group included 50 eyes of 25 patients, aged 40 to 81 years (mean 62.27 ± 10.81 years), with clinical cataract who were implanted with the Lumina accommodative IOL. The inclusion criteria of this study were as follows: patients with visual significant cataract with an expected positive effect of the surgery on the visual outcome. The patient had to be ≥ 40 years of age and with a calculated IOL power within the available diopter range. The exclusion criteria were comorbidities causing postoperative visual impairment such as degenerative macular pathology, glaucoma with optic disk damage and visual field loss, retinal dystrophies previous ocular surgeries such as vitrectomy , corneal graft surgery, lens subluxation or significant eye trauma that may induce lens instability, congenital ocular anomalies, endothelial cell count < 1200 cells/mm2 and previous known reading disabilities such as dyslexia. Only patients with less than 2 diopters (D) of corneal astigmatism were included in the study with no significant corneal irregularities (less than 0.5 microns of anterior corneal surface HOA) as measured by corneal topography (CSO, Costruzione Strumenti Oftalmici, Firenze, Italy). All patients were adequately informed and signed a consent form.

Preoperatively, all patients had a full ophthalmologic examination including the evaluation of the refractive status, keratometry, the distance and near visual acuities, slit lamp examination, applanation tonometry, and funduscopy. Distance and near visual acuity were measured with the ETDRS and the Radner reading chart (logarithm of reading acuity determination, logRAD), respectively. Other examinations included corneal topography Sirius/MS-39 (CSO, Costruzione Strumenti Oftalmici, Firenze, Italy), anterior segment optical coherence tomography MS-39 (CSO, Costruzione Strumenti Oftalmici, Firenze, Italy) or Casia2 (Tomey, Japan), posterior segment optical coherence tomography Cirrus OCT (Zeiss, Germany) and biometry IOL master 700 (Zeiss, Germany). The fixed optical power of the lens (i.e., the power required for an emmetropic eye) was calculated from optical biometry (IOL Master; Zeiss) by using proprietary Cþþ software integrated with Zemax ray-tracing software (Zemax, USA). The target refraction was plano in all cases that were included.

The same surgeon (JLA) performed all surgeries. All patients received retrobulbar anesthesia and mild sedation with midazolam. Adequate dilatation was obtained with intracameral mydriatics. The main corneal incision of 2.8 mm was placed temporally at the 180° meridian position in all eyes. A standard technique of phacoemulsification was performed followed by implantation of the Lumina in the sulcus plane of the eye by using a standard disposable injector system with an adapted, proprietary, AkkoLens butterfly cartridge. Postoperative topical therapy included a combination of topical antibiotics (ofloxacin 0.3%) and a steroid agent (dexamethasone 0.1%, Maxidex; Alcon, Spain).

The patients were evaluated during the follow up at five intervals: 1 day, 1 month, 3 months 6 months and a minimum of 12 months after surgery. In addition to the measurements listed in the preoperative protocol, the postoperative protocol included additional assessments of contrast sensitivity function in mesopic conditions (CSV 1000, VectorVision Ocular Health, Greenville, Ohio, USA) and the defocus curves. Monocular defocus curves were obtained with best distance refractive correction under low ambient light to keep an open pupil to minimize the undesirable effect of extended depth of focus owing to a small pupil, which can mask true accommodation. Negative and positive spherical lenses were added in 0.50 D steps, producing a stimulus for the eye to accommodate in the range from -5.00 to +2.00 D. The means of the measured visual acuities are summarized in mean defocus curves in which the measurements at 0.00 D and-2.50 D correspond to corrected distance visual acuity (CDVA) and corrected distance near visual acuity (CDNVA), respectively, and intermediate visual acuity corresponds to the measurement at -1.50 D. Depth of focus was evaluated from defocus curves at the levels of visual acuity of 0.10, 0.20, and 0.40 logMAR. The depth of focus for a particular eye was defined as the width of the defocus curve, in diopters, at a given level of visual acuity. The retinal optical quality was obtained using pyramidal aberrometry (Osiris, CSO, Italy) and optical quality analyzer system (OQAS, Visiomettrics SL, Spain) obtaining the MTF and PSF for different diameters and open field aberrometer (OFA, CSO, Italy) measured for distance and near.

Main outcome measures Primary: Distance and near visual acuities, defocus curve, accommodation, depth of focus.

Secondary: Contrast sensitivity function, optical quality assessment, PROMs (quality of vision and quality of life reported by the patients), complications.

ELIGIBILITY:
Inclusion Criteria:

* Visual significant cataract with an expected positive effect of the surgery on the visual outcome.
* ≥ 40 years of age
* Calculated IOL power within the available diopter range

Exclusion Criteria:

* Comorbidities causing postoperative visual impairment, such as degenerative macular pathology
* Glaucoma with optic disk damage and visual field loss
* Retinal dystrophies
* Previous ocular surgeries, such as vitrectomy, corneal graft surgery
* Lens subluxation
* Significant eye trauma that may induce lens instability
* Congenital ocular anomalies
* Endothelial cell count < 1200 cells/mm2
* Previous known reading disabilities, such as dyslexia.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Distance Vision measurements | minimum 12 months
  Distance and near visual acuities in LogMAR scale
Defocus curve measurements | minimum 12 months
  Defocus curve in diopters
Accommodation measurements | minimum 12 months
  Accommodation in diopters
Depth of focus measurements | minimum 12 months
  Depth of focus in diopters

SECONDARY OUTCOMES:
Contrast sensitivity function | minimum 12 months
  Contrast sensitivity function in cycles per degrees
Optical quality assessment | minimum 12 months
  Optical quality assessment in microns, PROMs (quality of vision and quality of life reported by the patients) considering a score from 1 (the best situation) to 5 (the worst situation)
Complications | minimum 12 months
  Complications not requiring units of measure

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alio, MD, PhD, Principal Investigator — Vissum Instituto Oftalmologico de Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alio JL, Simonov A, Plaza-Puche AB, Angelov A, Angelov Y, van Lawick W, Rombach M. Visual Outcomes and Accommodative Response of the Lumina Accommodative Intraocular Lens. Am J Ophthalmol. 2016 Apr;164:37-48. doi: 10.1016/j.ajo.2016.01.006. Epub 2016 Jan 29. PMID 26829595
- [Background] Alio JL, Simonov AN, Romero D, Angelov A, Angelov Y, van Lawick W, Rombach MC. Analysis of Accommodative Performance of a New Accommodative Intraocular Lens. J Refract Surg. 2018 Feb 1;34(2):78-83. doi: 10.3928/1081597X-20171205-01. PMID 29425385